CLINICAL TRIAL: NCT03083132
Title: Modafinil as a Novel Therapy for the Treatment of Freezing of Gait in Parkinson's Disease
Brief Title: Modafinil for Freezing of Gait (FOG) in Parkinson's Disease (PD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 206341
Record Dates: First submitted 2017-03-07; First posted 2017-03-17 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: freezing of gait
MeSH Terms: conditions — Parkinson Disease | interventions — Modafinil

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled delayed start
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Early-start (Active Comparator): 24 weeks of modafinil 50 mg oral daily
  Interventions: Drug: modafinil 50mg
- Delayed-start (Placebo Comparator): 12 weeks of oral placebo followed by 12 weeks of modafinil 50 mg oral daily
  Interventions: Drug: modafinil 50mg; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: modafinil 50mg — 1 capsule oral daily
Drug: Placebo oral capsule — 1 capsule oral daily
  Arms: Delayed-start

SUMMARY:
Freezing of gait is a late stage complication of Parkinson's disease in which patients note that their feet feel stuck or glued to the ground. This can lead to imbalance and falls and the secondary complications that can result from falls such as fractures and hospitalizations. While levodopa can help freezing of gait in some patients, it does not help in all, and the dose needed to treat freezing may be limited by side effects of the medications. Currently there are no treatments targeted towards freezing of gait and the goal of this research is to see if Modafinil could be one such drug to help freezing of gait in Parkinson's disease.

DETAILED DESCRIPTION:
Freezing of gait is a late stage complication of Parkinson's disease in which patients note that their feet feel stuck or glued to the ground. This can lead to imbalance and falls and the secondary complications that can result from falls such as fractures and hospitalizations. While levodopa can help freezing of gait in some patients, it does not help in all, and the dose needed to treat freezing may be limited by side effects of the medications. Currently there are no treatments targeted towards freezing of gait and the goal of this research is to see if Modafinil could be one such drug to help freezing of gait in Parkinson's disease.

Approximately 20 subjects aged 18 or older with idiopathic Parkinson's disease with freezing of gait will be asked to enroll in the study from the patient population in the movement disorders clinic at the University of Arkansas for Medical Sciences (UAMS). Subjects will be assigned randomly 1:1 to an early start and delayed start arm of the study. In the early start arm subjects will receive 24 weeks of 50 mg oral daily Modafinil while subjects in the delayed start arm will receive 12 weeks of placebo followed by 12 weeks of 50 mg oral daily Modafinil. Assessments will be performed prior to initiation of medication at the screening visit, as well as at 12 weeks of the treatment phase. The assessments will include questionnaires to determine the frequency and severity of freezing of gait, level of mood, anxiety and apathy and quality of life, physical examination and tests of cognitive function. Objective assessment of patients walking will be conducted using a pressure sensor impregnated mat at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD on UK brain bank criteria.
* Presence of FOG based on objective assessment by the movement disorders neurologist.
* FOG-Q score > 8.
* Stable PD therapy (including medications and stimulation) for a period of 3 months prior to trial enrollment.
* Age ≥ 50 years.

Exclusion Criteria:

* Patients on antidopaminergic medications for a period of less than 1 year from date of enrollment.
* Patients who may require adjustment of their PD medications over the 6 month period of the trial.
* History of allergic reactions to Modafinil or armodafinil.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, mitral valve prolapse, left ventricular hypertrophy, chronic obstructive pulmonary disease or psychiatric illness/social situations that would limit compliance with study requirements.
* Individuals who are pregnant or breastfeeding
* Non-english speaking individuals who are unable to complete the questionnaires and other assessments in English and/or follow instructions in English.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tuhin Virmani, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: First 12 Weeks (Placebo vs Modafinil)
Arm/Group | Early-start | Delayed-start
Started | 12 | 9
Completed | 12 | 7
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Last 12 Weeks (Drug for All Subjects)
Arm/Group | Early-start | Delayed-start
Started | 12 | 7
Completed | 11 | 6
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early-start | Delayed-start | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (6.3) | 72.9 (5.3) | 72.1 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 9 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 9 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21
Freezing of Gait Questionnaire (FOG-Q) [Mean (Standard Deviation); unit: units on a scale] — The freezing of gait questionnaire (FOG-Q) was administered by a movement disorders neurologist. The FOG-Q scores 6 items between 0 and 4, for a total score of 24; higher values indicate worse FOG.
  units on a scale | 13.8 (2.5) | 14.4 (1.7) | 14.0 (2.2)
Gait stride length (cm) [Mean (Standard Deviation); unit: cms] — Participants walked on a 20 foot instrumented gait mat for a total of 80 feet. The stride length was measured as the distance between two consecutive footsteps (for example right foot step to the next right footstep). The combined average stride length for both right and left feet are reported. Values usually range between 0 and 160 centimeters (the maximum stride length we have seen in an aging healthy population); lower values typically indicate more shuffling gait and have been associated with greater gait instability.
  cms | 69.8 (30.4) | 82.2 (27.3) | 75.1 (29.1)
motor Unified Parkinson's Disease Rating Scale (UPDRS) score [Mean (Standard Deviation); unit: units on a scale] — The motor Unified Parkinson's disease Rating scale (UPDRS) was administered by a movement disorders neurologist. The scale was administered in the levodopa-OFF state first at baseline (week 0), and again after taking the randomly assigned treatment (either Modafinil or placebo) for 12 weeks. The motor subscale of the UPDRS takes integer values between 0 and 4 for each of the 27 items for a total maximum score of 108; higher values indicate worse motor function.
  units on a scale | 37.7 (5.9) | 38.0 (8.3) | 37.8 (6.9)
Parkinson's Disease Questionnaire-39 (PDQ-39) [Mean (Standard Deviation); unit: units on a scale] — The Parkinson's Disease Questionnaire-39 (PDQ-39) was self-administered by participants. The PDQ-39 scores takes integer values between 0 and 4, for each of the 39 items for a total maximum score of 156; higher values indicate worse quality of life.
  units on a scale | 59.8 (21.1) | 60.7 (21.3) | 60.1 (20.7)
REM sleep Behavior Disorder Questionnaire (RBD-Q) [Mean (Standard Deviation); unit: units on a scale] — The REM sleep behavior disorder questionnaire (RBD-Q) was self administered by participants and measures the presence and severity of REM sleep behavior disorder. The RBD-Q maximum score is 13. Higher values indicate worse symptoms.
  units on a scale | 5.1 (3.5) | 5.3 (2.9) | 5.2 (3.2)
Epworth Sleepiness Scale (ESS) score [Mean (Standard Deviation); unit: units on a scale] — The Epworth Sleepiness Scale (ESS) was self administered by participants and measures the level of daytime sleepiness. The ESS maximum score is 24. Higher values indicate worse symptoms.
  units on a scale | 10.3 (2.9) | 10.1 (4.6) | 10.2 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline Freezing of Gait (FOG) After First 12 Weeks of Treatment, as Measured by the Giladi Freezing of Gait Questionnaire (FOG-Q).
Description: The freezing of gait questionnaire (FOG-Q) was administered by a movement disorders neurologist at baseline (week 0), and again after taking the randomly assigned treatment (either Modafinil or placebo) for 12 weeks. The FOG-Q scores 6 items between 0 and 4, for a total score of 24; higher values indicate worse FOG.
Time Frame: 12 weeks
Population: Participants that completed the placebo controlled portion of the study (first 12 weeks of the study)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early-start | Delayed-start
Number analyzed (Participants) | 12 | 7
units on a scale
  0 weeks (Baseline) | 13.75 (2.53) | 14.57 (1.62)
  12 weeks | 14.42 (4.03) | 13.43 (1.90)

2. Primary Outcome: Mean Change From Baseline Stride Length After 12 Weeks on Treatment, as Measured Using an Instrumented Gait Mat.
Description: Participants walked on a 20 foot instrumented gait mat for a total of 80 feet, first at baseline (week 0), and again after taking the randomly assigned treatment (either Modafinil or placebo) for 12 weeks. The stride length values usually range between 0 and 160 centimeters (the maximum stride length we have seen in an aging healthy population); lower values typically indicate more shuffling gait and have been associated with greater gait instability.
Time Frame: 12 weeks
Population: Participants that completed the placebo controlled portion of the study (first 12 weeks)
Measure: Mean (Standard Deviation); unit: cms
Arm/Group | Early-start | Delayed-start
Number analyzed (Participants) | 12 | 7
cms
  0 weeks (baseline) | 69.78 (30.37) | 90.13 (14.53)
  12 weeks | 64.04 (33.55) | 88.97 (15.91)

3. Secondary Outcome: Mean Change From Baseline in Motor Function After 12 Weeks on Treatment, as Measured by the Unified Parkinson's Disease Rating Scale Motor Score (UPDRS-III).
Description: For each participant, the Unified Parkinson's disease Rating scale (UPDRS) was administered by a movement disorders neurologist. The scale was first administered at baseline (week 0), and again after taking the randomly assigned treatment (either Modafinil or placebo) for 12 weeks. The motor subscale of the UPDRS takes integer values between 0 and 4 for each of the 27 items for a total maximum score of 108; higher values indicate worse motor function.
Time Frame: 12 weeks
Population: Subjects who completed the first 12 weeks of the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early-start | Delayed-start
Number analyzed (Participants) | 12 | 7
units on a scale
  0 weeks (baseline) | 37.71 (5.95) | 39.00 (9.11)
  12 weeks | 37.25 (10.02) | 34.36 (9.07)

4. Secondary Outcome: Mean Change From Baseline Quality of Life After 12 Weeks on Treatment, as Measured by the Parkinson's Disease Questionnaire-39 (PDQ-39).
Description: For each participant, the Parkinson's Disease Questionnaire (PDQ-39) was self-administered by participants. The questionnaire was first administered at baseline (week 0), and again after taking the randomly assigned treatment (either Modafinil or placebo) for 12 weeks. The PDQ-39 scores takes integer values between 0 and 4, for each of the 39 items for a total maximum score of 156; higher values indicate worse quality of life.
Time Frame: 12 weeks
Population: Participants that completed the placebo controlled portion of the study (first 12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early-start | Delayed-start
Number analyzed (Participants) | 12 | 7
units on a scale
  0 weeks (baseline) | 59.8 (21.1) | 65.7 (21.2)
  12 weeks | 62.6 (17.5) | 63.3 (23.5)

5. Secondary Outcome: Mean Change From Baseline Sleep Quality After 12 Weeks on Treatment, as Measured by the REM Sleep Behavior Disorder Questionnaire (RBD-Q).
Description: For each participant, the REM sleep behavior disorder questionnaire (RBD-Q) was self-administered by participants. The questionnaires were first administered at baseline (week 0), and again after taking the randomly assigned treatment (either Modafinil or placebo) for 12 weeks. The RBD-Q score takes integer values between 0 and 1, for each of the 13 item yes/no questions for a total maximum score of 13; higher values indicate worse sleep behavior disorder.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early-start | Delayed-start
Number analyzed (Participants) | 12 | 7
units on a scale
  0 weeks (baseline) | 5.08 (3.53) | 5.42 (2.37)
  12 weeks | 5.58 (3.65) | 3.57 (2.37)

6. Secondary Outcome: Mean Change From Baseline Sleep Quality After 12 Weeks on Treatment, as Measured by the Epworth Sleepiness Scale (ESS).
Description: For each participant, the Epworth Sleepiness Scale (ESS) questionnaires was self-administered by participants. The questionnaires were first administered at baseline (week 0), and again after taking the randomly assigned treatment (either Modafinil or placebo) for 12 weeks. The ESS takes integer values between 0 and 3, for each of the 8 items for a total maximum score of 24; higher values indicate more daytime sleepiness.
Time Frame: 12 weeks
Population: Participants that completed the placebo controlled portion of the study (first 12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early-start | Delayed-start
Number analyzed (Participants) | 12 | 7
units on a scale
  0 weeks (baseline) | 10.33 (2.90) | 9.00 (4.58)
  12 weeks | 10.25 (4.35) | 8.71 (2.69)

ADVERSE EVENTS:
Time Frame: Period of the trial (30 weeks)
Arm/Group | Early-start | Delayed-start
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/9
Other Adverse Events (participants affected / at risk) | 12/12 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early-start (N=12) | Delayed-start (N=9)
Cervical stenosis (Nervous system disorders) | 1 (1) | 0 (0) — Participant was diagnosed with cervical stenosis during the course of the trial and underwent surgical procedure. As a result it was determined appropriate for him to discontinue further study assessments.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early-start (N=12) | Delayed-start (N=9)
lower extremity edema (Cardiac disorders) | 0 | 1
dyspnea on exertion (Cardiac disorders) | 0 | 1
palpitations (Cardiac disorders) | 0 | 1
lightheadedness on standing (Cardiac disorders) | 1 | 0
dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
facial rash (Skin and subcutaneous tissue disorders) | 1 | 0
skin tag (Skin and subcutaneous tissue disorders) | 1 | 0
cold intolerance (Endocrine disorders) | 0 | 1
diagnosed with diabetes (Endocrine disorders) | 1 | 0
rhinorrhea (General disorders) | 2 | 2
allergy flare (General disorders) | 0 | 1
lower eyelid edema (Eye disorders) | 1 | 0
tinnitus (Ear and labyrinth disorders) | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 1
constipation (Gastrointestinal disorders) | 0 | 1
hyperphagia (Metabolism and nutrition disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 1 | 0
calf pain/cramps (Musculoskeletal and connective tissue disorders) | 2 | 2
bursitis/epicondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
neck stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
paresthesias (Nervous system disorders) | 1 | 1
morning grogginess (Nervous system disorders) | 0 | 1
daytime sleepiness (Nervous system disorders) | 1 | 1
insomnia (Nervous system disorders) | 1 | 3
falls (Nervous system disorders) | 1 | 2
sciatica (Nervous system disorders) | 0 | 1
daytime confusion (Nervous system disorders) | 1 | 0
dysphagia (Nervous system disorders) | 1 | 0
fatigue (Nervous system disorders) | 1 | 0
hallucinations (Nervous system disorders) | 1 | 0
hand cramps (Nervous system disorders) | 1 | 0
freezing of gait (Nervous system disorders) | 1 | 0
headaches (Nervous system disorders) | 2 | 1
imbalance (Nervous system disorders) | 2 | 0
difficulty getting out of bed (Nervous system disorders) | 1 | 0
difficulty with ADLs (Nervous system disorders) | 1 | 0
slowed gait (Nervous system disorders) | 1 | 0
toe walking (Nervous system disorders) | 1 | 0
word finding difficulty (Nervous system disorders) | 1 | 0
lacrimation (Eye disorders) | 1 | 1
visual floaters/flashing (Eye disorders) | 1 | 1
blurred vision (Eye disorders) | 1 | 0
anxiety (Psychiatric disorders) | 1 | 2
depressed mood (Psychiatric disorders) | 1 | 0
irritability (Psychiatric disorders) | 1 | 0
nocturia (Renal and urinary disorders) | 4 | 1
nephrolithiasis (Renal and urinary disorders) | 1 | 0
urinary incontinance (Renal and urinary disorders) | 1 | 0
urinary tract infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT03083132/Prot_SAP_001.pdf